CLINICAL TRIAL: NCT05565976
Title: Dapagliflozin Effect in Cognitive Impairment in Stroke Trial
Acronym: DECIST
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jaime Daniel Mondragon (Other)
Collaborators: Hospital General León (Unknown); Hospital General de Zona IMSS N0. 21 (Unknown); University Medical Center Groningen (Other)
Responsible Party: Sponsor-Investigator, Jaime Daniel Mondragon, Principal Investigator, Clinical Professor, Universidad de Guanajuato
Organization: Universidad de Guanajuato (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: F-2022-1005-016
Record Dates: First submitted 2022-09-20; First posted 2022-10-04 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2022-10

CONDITIONS: Stroke, Ischemic; Mild Cognitive Impairment; Dementia, Vascular; Metabolic Syndrome
Keywords: dapagliflozin; mortality; cognitive impairment
MeSH Terms: conditions — Ischemic Stroke; Cognitive Dysfunction; Dementia, Vascular; Metabolic Syndrome | interventions — dapagliflozin; Hydroxymethylglutaryl-CoA Reductase Inhibitors; Cardiovascular Agents; Atorvastatin; Pravastatin; Rosuvastatin Calcium; Platelet Aggregation Inhibitors; Clopidogrel; Aspirin; Hypoglycemic Agents; Sulfonylurea Compounds; meglitinide; Biguanides; Thiazolidinediones; Bromocriptine; Insulin Glargine; Insulin Lispro; Insulin, Isophane

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Duoble-blinded study, only outcome assessor will have knowledge of labels.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Dapagliflozin (Experimental): 10mg PO q24h for 12 months plus standard treatment with statins, platelet antiaggregant, and hypoglycemic medications.
  Interventions: Drug: Dapagliflozin 10mg Tab; Drug: Statins (Cardiovascular Agents); Drug: Platelet Antiaggregant; Drug: Antidiabetic
- Standard treatment (Active Comparator): Standard treatment with statins, platelet antiaggregant, and hypoglycemic medications.
  Interventions: Drug: Statins (Cardiovascular Agents); Drug: Platelet Antiaggregant; Drug: Antidiabetic

INTERVENTIONS:
Drug: Dapagliflozin 10mg Tab — 10mg PO q24h for 12 months
  Other Names: FORXIGA
  Arms: Dapagliflozin
Drug: Statins (Cardiovascular Agents) — Atorvastatin 20mg PO q24h or Pravastatin 20mg PO q24h or Rosuvastatin 10mg PO q24h
  Other Names: Atorvastatin; Pravastatin; Rosuvastatin
Drug: Platelet Antiaggregant — Clopidogrel 75mg PO q24h or Acetylsalicylic acid 100mg PO q24h
  Other Names: Clopidogrel; Acetylsalicylic acid
Drug: Antidiabetic — Previously established medical treatment for type 2 diabetes will be maintained.
  Other Names: Sulfonylureas; Meglitinides; Biguanides; Thiazolidinediones; α-Glucosidase inhibitors; Inhibitors of dipeptidyl peptidase 4; Cycloset; Insulin glargine; Insulin lispro; Isophane insulin

SUMMARY:
Background: Dementia is an international public health problem, affecting approximately 50,000,000 people worldwide in 2018 and will triple by 2050; furthermore, reaching an approximate cost of 4 billion dollars. Given its high worldwide prevalence and probable underdiagnosis, the international guidelines for the assessment of dementia syndromes recommend the assessment of cognitive impairment in patients over 55 years of age as part of clinical practice in patients who presented an ischemic cerebrovascular event. Several risk factors associated with cognitive impairment in cerebrovascular disease are identified in the literature: 1) demographic factors (e.g., age over 65 years and female sex); 2) risk factors present prior to the ischemic stroke (e.g., cognitive impairment, physical impairment); 3) factors utilized to assess the severity of an ischemic stroke (e.g., supratentorial location, ischemic stroke in the dominant hemisphere, recurrence of ischemic strokes); 4) post-ischemic stroke factors (e.g., delirium and seizures); and 5) factors associated with neuroimaging findings (e.g., cerebral small vessel disease, cortical atrophy, and medial temporal lobe atrophy).

This is a randomized controlled trial in individuals with an acute ischemic stroke without dementia that will be treated with 10mg dapagliflozin PO q24h for 12 months and standard treatment against only standard treatment (i.e., statins, platelet antiaggregant, and hypoglycemic medications) when appropriate. The outcome measure evaluated will be global cognitive function. Cardiovascular risk factors will be associated with cognitive decline.

DETAILED DESCRIPTION:
Detailed Description: This is a double-blind, randomized, placebo-controlled, parallel-group, 12-month longitudinal study performed at a single center (Hospital General de Zona con Medicina Familiar IMSS No. 21, León Guanajuato, México) designed to investigate the effect of dapagliflozin in participants with a recent acute stroke but no history of dementia (CDR score ≤ 0.5). A total of 270 participants are to be included (i.e., 135 on each arm).

Overall objective: To assess the effect of Dapagliflozin on cardiovascular risk (i.e., the volume of epicardial fat, volume of total carotid atherosclerotic plaque, and coronary artery calcium score) in patients with ischemic cerebrovascular disease dependent on global cognitive function at a second level teaching hospital in Mexico.

Statistical analysis: Descriptive statistics will be reported for all included variables. Statistical analysis will be performed using SPSS 25 (SPSS Inc., Chicago, IL). All variables will be examined to determine the existence of outliers and whether they meet the assumptions about a Gaussian distribution. The Shapiro-Wilk tests will be used to determine normality distribution, as well as visual inspection of histograms and Q-Q plots. Demographic and clinical variables will be summarized in proportions and percentages. The categorical variables will be evaluated to determine statistical inferences with the Mann-Whitney U test. Continuous variables will be assessed for statistical inferences using t-tests (e.g., simple, paired, one, and two samples) and Levene's test to assess equality of variances. The Kaplan-Meier method will be used to calculate the distributions of mortality and development of mild amnestic cognitive disorder and dementia syndrome. The Gehan-Breslow-Wilcoxon method will be used to assess the equality of the mortality distributions and the development of mild amnestic cognitive disorder or dementia syndrome. A multivariate analysis will be performed with a Cox regression model to assess the variables that predict mortality, and the development of a mild amnestic cognitive disorder, or dementia syndrome at 6 and 12 months in case there are differences in mortality distributions. Statistical significance will be set at p=0.05 and a Bonferroni correction will be performed for multiple comparisons.

ELIGIBILITY:
Inclusion Criteria:

* Ages of 60 and 80 years
* Both sexes
* Cerebrovascular ischemic event within 15 days
* Clinical dementia rating score ≤ 0.5
* Signed informed consent

Exclusion Criteria:

* Type 1 diabetes mellitus
* Aphasia
* Incomplete neuropsychological battery
* Previously diagnosed dementia
* Cerebrovascular ischemic stroke older than 15 days
* History of hemorrhagic cerebrovascular event
* Neoplasia diagnosis or evidence of a metastatic process, glomerular filtration rate < 45 mL/min at the time of inclusion
* Liver enzyme test alterations (i.e., aspartate transaminase or alanine transaminase three times greater than normal levels, total bilirubin> 2.0 mg/dL
* Previously taking SGLT2 inhibitors
* History of diabetic ketoacidosis
* Recurrent urinary tract infections
* Psychiatric disorders (e.g., dementia, psychosis, bipolar disorder, among others).
* Less than a 12-month follow-up
* Inability to perform chest CT (e.g., claustrophobia)
* Incomplete medical files pertaining to the variables of interest
* Less than 12-month follow-up
* Decision to withdraw their participation at any moment
* Poor adherence to medical treatment
* Reported and documented disease complications or adverse effects (e.g., severe glycemic imbalance, diabetic ketoacidosis, or hyperosmolar hyperglycemic state, altered hepatic enzyme tests)

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Change in Clinical Dementia Rating score as a proxy of cognitive deterioration | 6 and 12 months
  Time-to-event analysis using the Kaplan-meier survival analysis via increase in Clinical Dementia Rating score greter or equal to 0.5

SECONDARY OUTCOMES:
Number of strokes after initial cerebrovascular event | 12 months
  Independent stroke events

OTHER OUTCOMES:
Adverse effects due to Dapagliflozin | 12 months
  Adverse effects reported due to the use of dapagliflozin

CONTACTS AND LOCATIONS:
Overall Officials: Gabriela G López-Hernández, M.D., Study Chair — Hospital General de Zona IMSS 21; Lizeth C Ramírez-Zamudio, M.D., Study Chair — Hospital General de Zona IMSS 21; Jaime D Mondragón, M.D., Ph.D., Principal Investigator — University Medical Center Groningen, Department of Neurology, Alzheimer Center Groningen
Locations (1):
- Hospital General de Zona IMSS 21, León, Guanajuato, Mexico

IPD SHARING:
Plan to Share IPD: Yes
The study protocol, statistical analysis plan and informed consent form are available through the IMSS platform or upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Starting august 2022
Access Criteria: Request IMSS institutional board

REFERENCES:
- [Result] Bjergfelt SS, Sorensen IMH, Hjortkjaer HO, Landler N, Ballegaard ELF, Biering-Sorensen T, Kofoed KF, Lange T, Feldt-Rasmussen B, Sillesen H, Christoffersen C, Bro S. Carotid plaque thickness is increased in chronic kidney disease and associated with carotid and coronary calcification. PLoS One. 2021 Nov 23;16(11):e0260417. doi: 10.1371/journal.pone.0260417. eCollection 2021. PMID 34813630
- [Result] Cherney DZI, Dekkers CCJ, Barbour SJ, Cattran D, Abdul Gafor AH, Greasley PJ, Laverman GD, Lim SK, Di Tanna GL, Reich HN, Vervloet MG, Wong MG, Gansevoort RT, Heerspink HJL; DIAMOND investigators. Effects of the SGLT2 inhibitor dapagliflozin on proteinuria in non-diabetic patients with chronic kidney disease (DIAMOND): a randomised, double-blind, crossover trial. Lancet Diabetes Endocrinol. 2020 Jul;8(7):582-593. doi: 10.1016/S2213-8587(20)30162-5. PMID 32559474
- [Result] Dekkers CCJ, Petrykiv S, Laverman GD, Cherney DZ, Gansevoort RT, Heerspink HJL. Effects of the SGLT-2 inhibitor dapagliflozin on glomerular and tubular injury markers. Diabetes Obes Metab. 2018 Aug;20(8):1988-1993. doi: 10.1111/dom.13301. Epub 2018 Apr 23. PMID 29573529
- [Result] Dhillon S. Dapagliflozin: A Review in Type 2 Diabetes. Drugs. 2019 Jul;79(10):1135-1146. doi: 10.1007/s40265-019-01148-3. PMID 31236801
- [Result] Diaz-Rodriguez E, Agra RM, Fernandez AL, Adrio B, Garcia-Caballero T, Gonzalez-Juanatey JR, Eiras S. Effects of dapagliflozin on human epicardial adipose tissue: modulation of insulin resistance, inflammatory chemokine production, and differentiation ability. Cardiovasc Res. 2018 Feb 1;114(2):336-346. doi: 10.1093/cvr/cvx186. PMID 29016744
- [Result] Esterline R, Oscarsson J, Burns J. A role for sodium glucose cotransporter 2 inhibitors (SGLT2is) in the treatment of Alzheimer's disease? Int Rev Neurobiol. 2020;155:113-140. doi: 10.1016/bs.irn.2020.03.018. Epub 2020 Aug 11. PMID 32854852
- [Result] Esterline RL, Vaag A, Oscarsson J, Vora J. MECHANISMS IN ENDOCRINOLOGY: SGLT2 inhibitors: clinical benefits by restoration of normal diurnal metabolism? Eur J Endocrinol. 2018 Apr;178(4):R113-R125. doi: 10.1530/EJE-17-0832. Epub 2018 Jan 25. PMID 29371333
- [Result] Fani L, van Dam-Nolen DHK, Vernooij M, Kavousi M, van der Lugt A, Bos D. Circulatory markers of immunity and carotid atherosclerotic plaque. Atherosclerosis. 2021 May;325:69-74. doi: 10.1016/j.atherosclerosis.2021.03.040. Epub 2021 Apr 7. PMID 33894597
- [Result] Iacobellis G, Gra-Menendez S. Effects of Dapagliflozin on Epicardial Fat Thickness in Patients with Type 2 Diabetes and Obesity. Obesity (Silver Spring). 2020 Jun;28(6):1068-1074. doi: 10.1002/oby.22798. Epub 2020 Apr 30. PMID 32352644
- [Result] Iadecola C, Duering M, Hachinski V, Joutel A, Pendlebury ST, Schneider JA, Dichgans M. Vascular Cognitive Impairment and Dementia: JACC Scientific Expert Panel. J Am Coll Cardiol. 2019 Jul 2;73(25):3326-3344. doi: 10.1016/j.jacc.2019.04.034. PMID 31248555
- [Result] Ihara M, Saito S. Drug Repositioning for Alzheimer's Disease: Finding Hidden Clues in Old Drugs. J Alzheimers Dis. 2020;74(4):1013-1028. doi: 10.3233/JAD-200049. PMID 32144994
- [Result] Jabbour S, Seufert J, Scheen A, Bailey CJ, Karup C, Langkilde AM. Dapagliflozin in patients with type 2 diabetes mellitus: A pooled analysis of safety data from phase IIb/III clinical trials. Diabetes Obes Metab. 2018 Mar;20(3):620-628. doi: 10.1111/dom.13124. Epub 2017 Oct 26. PMID 28950419
- [Result] Jellinger KA, Attems J. Prevalence of dementia disorders in the oldest-old: an autopsy study. Acta Neuropathol. 2010 Apr;119(4):421-33. doi: 10.1007/s00401-010-0654-5. Epub 2010 Mar 4. PMID 20204386
- [Result] McMurray JJV, Solomon SD, Inzucchi SE, Kober L, Kosiborod MN, Martinez FA, Ponikowski P, Sabatine MS, Anand IS, Belohlavek J, Bohm M, Chiang CE, Chopra VK, de Boer RA, Desai AS, Diez M, Drozdz J, Dukat A, Ge J, Howlett JG, Katova T, Kitakaze M, Ljungman CEA, Merkely B, Nicolau JC, O'Meara E, Petrie MC, Vinh PN, Schou M, Tereshchenko S, Verma S, Held C, DeMets DL, Docherty KF, Jhund PS, Bengtsson O, Sjostrand M, Langkilde AM; DAPA-HF Trial Committees and Investigators. Dapagliflozin in Patients with Heart Failure and Reduced Ejection Fraction. N Engl J Med. 2019 Nov 21;381(21):1995-2008. doi: 10.1056/NEJMoa1911303. Epub 2019 Sep 19. PMID 31535829
- [Result] Mijajlovic MD, Pavlovic A, Brainin M, Heiss WD, Quinn TJ, Ihle-Hansen HB, Hermann DM, Assayag EB, Richard E, Thiel A, Kliper E, Shin YI, Kim YH, Choi S, Jung S, Lee YB, Sinanovic O, Levine DA, Schlesinger I, Mead G, Milosevic V, Leys D, Hagberg G, Ursin MH, Teuschl Y, Prokopenko S, Mozheyko E, Bezdenezhnykh A, Matz K, Aleksic V, Muresanu D, Korczyn AD, Bornstein NM. Post-stroke dementia - a comprehensive review. BMC Med. 2017 Jan 18;15(1):11. doi: 10.1186/s12916-017-0779-7. PMID 28095900
- [Result] Mohamed Fuad Z, Mahadzir H, Syed Zakaria SZ, Mohamed Ibrahim N. Frequency of Cognitive Impairment Among Malaysian Elderly Patients Following First Ischaemic Stroke-A Case Control Study. Front Public Health. 2020 Nov 12;8:577940. doi: 10.3389/fpubh.2020.577940. eCollection 2020. PMID 33282811
- [Result] Sato T, Aizawa Y, Yuasa S, Fujita S, Ikeda Y, Okabe M. The Effect of Dapagliflozin Treatment on Epicardial Adipose Tissue Volume and P-Wave Indices: An Ad-hoc Analysis of The Previous Randomized Clinical Trial. J Atheroscler Thromb. 2020 Dec 1;27(12):1348-1358. doi: 10.5551/jat.48009. Epub 2020 Feb 28. PMID 32115470
- [Result] Serena J, Irimia P, Calleja S, Blanco M, Vivancos J, Ayo-Martin O; Representacion de la Sociedad Espanola de Neurosonologia (SONES). [Ultrasound measurement of carotid stenosis: recommendations from the Spanish Society of Neurosonology]. Neurologia. 2013 Sep;28(7):435-42. doi: 10.1016/j.nrl.2012.07.011. Epub 2012 Oct 4. Spanish. PMID 23040716
- [Result] Suda S, Nishimura T, Ishiwata A, Muraga K, Aoki J, Kanamaru T, Suzuki K, Sakamoto Y, Katano T, Nishiyama Y, Mishina M, Kimura K. Early Cognitive Impairment after Minor Stroke: Associated Factors and Functional Outcome. J Stroke Cerebrovasc Dis. 2020 May;29(5):104749. doi: 10.1016/j.jstrokecerebrovasdis.2020.104749. Epub 2020 Mar 14. PMID 32178931
- [Result] Uemura MT, Maki T, Ihara M, Lee VMY, Trojanowski JQ. Brain Microvascular Pericytes in Vascular Cognitive Impairment and Dementia. Front Aging Neurosci. 2020 Apr 14;12:80. doi: 10.3389/fnagi.2020.00080. eCollection 2020. PMID 32317958
- [Result] van der Flier WM, Skoog I, Schneider JA, Pantoni L, Mok V, Chen CLH, Scheltens P. Vascular cognitive impairment. Nat Rev Dis Primers. 2018 Feb 15;4:18003. doi: 10.1038/nrdp.2018.3. PMID 29446769
- [Result] Zlokovic BV, Gottesman RF, Bernstein KE, Seshadri S, McKee A, Snyder H, Greenberg SM, Yaffe K, Schaffer CB, Yuan C, Hughes TM, Daemen MJ, Williamson JD, Gonzalez HM, Schneider J, Wellington CL, Katusic ZS, Stoeckel L, Koenig JI, Corriveau RA, Fine L, Galis ZS, Reis J, Wright JD, Chen J. Vascular contributions to cognitive impairment and dementia (VCID): A report from the 2018 National Heart, Lung, and Blood Institute and National Institute of Neurological Disorders and Stroke Workshop. Alzheimers Dement. 2020 Dec;16(12):1714-1733. doi: 10.1002/alz.12157. Epub 2020 Oct 8. PMID 33030307